CLINICAL TRIAL: NCT07178873
Title: Effects of a Psychosocial Teleassistance Programme for Adults With Spina Bifida
Brief Title: Psychosocial Teleassistance Programme for Adults With Spina Bifida
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuro-e-Motion SB
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Spina Bifida; Self Esteem; Quality of Life (QOL); Self Concept; Anxiety; Depression; Interpersonal Needs
MeSH Terms: conditions — Spinal Dysraphism; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial teleassistance intervention (Experimental): Psychosocial intervention, comprising 10 group sessions, followed by two 3-month follow-up sessions, is offered.
  Interventions: Behavioral: Psychosocial teleassistance intervention
- Wait list (Experimental): Waiting list control group.
  Interventions: Behavioral: Psychosocial teleassistance intervention

INTERVENTIONS:
Behavioral: Psychosocial teleassistance intervention — The teleassistance psychosocial intervention involves 10 weekly 90-minute group sessions, with each group comprising 6 to 7 participants. These sessions are designed to enhance self-concept, self-esteem and social skills, reduce symptoms, and improve overall psychological well-being. Two follow-up sessions will be provided three months after the main program concludes.

SUMMARY:
This clinical trial assesses the effect of a telecare psychosocial intervention designed for adults with spina bifida. The intervention consists of 10 weekly 1.5-hour group sessions, followed by two 3-month follow-up sessions. Each group will consist of 6 to 7 individuals. The intervention is aimed at strengthening aspects of self-concept, self-esteem, social skills and aims at a reduction of symptomatology and a general improvement of psychological well-being.

DETAILED DESCRIPTION:
The present study undertakes the development and evaluation of a structured, psychosocial teleassistance intervention designed for adult individuals with spina bifida. The variables of interest and intervention include quality of life, self-esteem, self-concept, anxious-depressive symptomatology, interpersonal needs and coping strategies. The study aims to test whether the psychosocial teleassistance programme improves the aforementioned variables.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with spina bifida by a specialist.
* Being between 18 and 75 years old.
* Having their informed consent or the informed consent of their legal guardians.
* Having Spanish as one of their main languages.
* Having access to a computer (with a camera, microphone and speakers integrated) and Internet connection to take part in the videoconferences.

Exclusion Criteria:

* Age that is inconsistent with the established range.
* The presence of any comorbid diagnosis or sensory deficit that would impede the effective execution of the intervention's activities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life - The World Health Organization WHOQOL-BREF Quality of Life Assessment | 3 months after the intervention
  The World Health Organization WHOQOL-BREF Quality of Life Assessment (WHOQOL-BREF) is a tool designed to assess quality of life using twenty-six items. The questionnaire measures four different domains: physical health, psychological health, social relationships, and environment. Domain scores are transformed to a scale ranging from 0 to 100. Higher scores reflect better quality of life.
Anxiety and depression - The Hospital Anxiety and Depression Scale | 3 months after the intervention
  The Hospital Anxiety and Depression Scale (HADS) is a scale primarily designed to assess anxiety and depressive symptomatology using 14 items. The instrument is composed of two subscales: an anxiety subscale and a depression subscale. Total scores on each subscale range from 0 to 21, where a higher score is indicative of greater symptom severity.
Depression - The Patient Health Questionnaire | 3 months after the intervention
  The Patient Health Questionnaire (PHQ-9) is a brief, nine-item tool designed to detect and measure the severity of depression. The score can range from 0 to 27. Higher scores reflect more severe depressive symptoms, whereas lower scores indicate minimal or no depressive symptoms.
Self-esteem - The Rosenberg Self-Esteem Scale | 3 months after the intervention
  The Rosenberg Self-Esteem Scale (RSE) is a 10-item scale designed to assess self-esteem. The final score ranges from 10 to 40. Higher scores reflect greater self-esteem, whereas lower scores indicate reduced self-esteem.
Self-Concept - Self-Concept Questionnaire Form-5 | 3 months after the intervention
  The Self-Concept Questionnaire Form-5 (AF-5) is an instrument used to evaluate self-concept across five dimensions: social, academic-work/professional, emotional, family, and physical. Domain scores are transformed to a scale ranging from 0 to 10. Higher scores indicate a better self-concept across domains, while lower scores reflect worse self-concept in those areas.

SECONDARY OUTCOMES:
Functionality - The Barthel Index | 3 months after the intervention
  The Barthel Index (IB) is an instrument used to evaluate physical functionality and level of independence across ten basic activities of daily living. Scores range from 0 to 100. A higher score reflects better functional independence, whereas a lower score indicates greater dependence for daily activities.
Coping strategies - The Brief Cope Stress Questionnaire | 3 months after the intervention
  The Brief Cope Stress Questionnaire (COPE-28) is an instrument that consists of 28 items used to assess fourteen coping strategies: active coping, planning, instrumental support, emotional support, self-distraction, venting, disengagement, positive reinterpretation, denial, acceptance, religion, substance use, humor, and self-blame. Higher scores indicate greater use of specific coping strategies, while lower scores reflect less frequent use.
Interpersonal Needs - The Interpersonal Needs Questionnaire | 3 months after the intervention
  The Interpersonal Needs Questionnaire (INQ) is designed to assess the degree of frustration with various interpersonal needs. This 12-item questionnaire is divided into two subscales: thwarted belongingness and perceived burdensomeness. Higher scores reflect higher levels of perceived burdensomeness and thwarted belongingness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Deusto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The plan is open for other researchers to contact the principal investigator of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is available from now until 2027.
Access Criteria: The plan is open for other researchers to contact the principal investigator of the study.

REFERENCES:
- [Background] Ordoñez-Carrasco, J. L., Salgueiro, M., Sayans-Jiménez, P., Blanc-Molina, A., García-Leiva, J. M., Calandre, E. P. y Rojas, A. J. Propiedades psicométricas de la versión en español del Cuestionario de Necesidades Interpersonales de 12 ítems en pacientes con síndrome de fibromialgia. Anales de Psicología. 2018; 34(2), 274-282. https://doi.org/10.6018/analesps.34.2.293101
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Background] García, F. y Musitu, G. (1999). Autoconcepto Forma 5 (AF5). TEA Ediciones.
- [Background] Baztán, J. J., Pérez del Molino, J., Alarcón, T., San Cristóbal, E., Izquierdo, G. y Manzabeitia, J. Índice de Barthel: instrumento válido para la valoración funcional de pacientes con enfermedad cerebrovascular. Revista Española de Geriatría y Gerontología. 1993; 28(1), 32-40.
- [Background] Morán, C., Landero, R. y González, M. T. COPE-28: un análisis psicométrico de la versión en español del Brief COPE. Universitas Psychologica. 2010; 9(2), 543-552.
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Fernández-Montalvo, J. y Echeburúa, E. Variables psicopatológicas y distorsiones cognitivas de los maltratadores en el hogar: Un análisis descriptivo. Análisis y Modificación de Conducta. 1997; 23(88), 151-180.
- [Background] Rosenberg, A. (1965). Society and the adolescent self-image. Princenton.
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] López-Roig, S., Terol, M.C., Pastor, M.A., Neipp, M.C., Massutí, B., Rodríguez-Marín. J., Leyda, J.I., Martín-Aragón, M. y Sitges, E. Ansiedad y Depresión. Validación de la escala HAD en pacientes oncológicos. Revista de Psicología de la Salud. 2000; 12(2): 127-155. doi.org/10.21134/pssa.v12i2.787
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Lucas-Carrasco R. The WHO quality of life (WHOQOL) questionnaire: Spanish development and validation studies. Qual Life Res. 2012 Feb;21(1):161-5. doi: 10.1007/s11136-011-9926-3. Epub 2011 May 25. PMID 21611868
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712